CLINICAL TRIAL: NCT05756894
Title: Pilot Study: Spike-timing-dependent Plasticity for Respiratory Function After Spinal Cord Injury
Brief Title: Neurostimulation for Respiratory Function After Spinal Cord Injury
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shirley Ryan AbilityLab (Other)
Responsible Party: Principal Investigator, Monica Perez, Scientific Chair, Arms and Hands Lab, Shirley Ryan AbilityLab
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU00217043
Record Dates: First submitted 2023-02-23; First posted 2023-03-07 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Spinal Cord Injuries; Cervical Spinal Cord Injury; Respiratory Function Impaired
Keywords: Neural plasticity; Spinal cord injury; Diaphragm; Respiratory training; Spike-timing-dependent plasticity; Neurostimulation
MeSH Terms: conditions — Spinal Cord Injuries; Respiratory Insufficiency

STUDY DESIGN:
Intervention Model Description: Participants with high cervical spinal cord injury will receive 40 treatment sessions (STDP stimulation and respiratory training) and will be asked to complete pre-, Post-20, and Post-40 assessment sessions.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Neurostimulation for respiratory function after spinal cord injury (Experimental): Efficacy of STDP on respiratory function.
  Interventions: Device: Neurostimulation; Other: Repiratory training

INTERVENTIONS:
Device: Neurostimulation — Paired stimulation will be given to the spinal cord and to peripheral nerves so that the signals are received at the spinal cord at a specific interval.
  Other Names: Spike-timing-dependent plasticity (STDP stimulation); Neural plasticity
Other: Repiratory training — Respiratory exercises will be completed immediately after completing neurostimulation. Respiratory exercises will involve inspiratory muscle training performing four sets of 6-10 breaths per day with two minutes of rest.

SUMMARY:
The purpose of this research study is to learn more about the connections between the brain, nerves, and diaphragm after experiencing a cervical spinal cord injury (SCI).The main question it aims to answer is:

Changes in respiratory function and recovery using stimulation and respiratory exercise training in spinal cord-injured individuals.

Participants will complete a maximum of 55 study visits. They will be asked to complete about 40 treatment sessions which include multiple stimulation sessions over the scalp and neck, followed by about 60 minutes of respiratory training. Assessment sessions will be completed prior at baseline, after 20 sessions and after 40 sessions of study treatment.

DETAILED DESCRIPTION:
The purpose of this study is to test a strategy to potentiate functional recovery of respiratory function in individuals with spinal cord injury (SCI). Respiratory function is often impaired in individuals with high cervical spinal cord injury (SCI, C1-C5) leading to reduced quality of life and mortality. Currently, research has shown Spike-timing-dependent plasticity (STDP) targeting cortico-motoneuronal connections effectively promote recovery in upper and lower limbs, including functions such as grasping and locomotion. The overall goal of our proposal is to develop a non-invasive protocol using

STDP that can be used to strengthen synaptic plasticity and voluntary motor output in the diaphragm muscle in humans with high cervical SCI. To assess the effect of STDP on respiratory function in humans with high cervical SCI, we propose a pilot study of efficacy trial with the specific aim below:

The overall objective of this project is to investigate the efficacy of spike-timing-dependent plasticity (STDP) on respiratory function in humans with high cervical SCI.

Specific Aim: Examine the effect of STDP in respiratory function in humans with chronic high cervical SCI.

ELIGIBILITY:
Inclusion Criteria:

1. Male and females between ages 18-85 years
2. SCI at least 6 months post-injury
3. Spinal Cord injury at C1-C5
4. Demonstrate respiratory deficit following spinal cord injury as following: (1) Individuals using mechanical ventilation, and (2) individuals with pulmonary function testing (PFT) deficits corresponding to having a vital capacity (VC) < 80% (predicted)
5. Must have a family member or caregiver who is trained and willing to operate the mechanical ventilator during study visits.

Exclusion Criteria:

1. Any illness or condition that based on the research team's assessment, will compromise with the participant's ability to comply with the protocol, patient safety, or the validity of the data collected during this study.
2. Any debilitating disease prior to the SCI that caused exercise intolerance.
3. Individuals entirely dependent on the support of a diaphragmatic pacer (24 hours per day).
4. Premorbid, ongoing major depression or psychosis, altered cognitive status.
5. History of head injury or stroke
6. Vascular, traumatic, tumoral, infectious, or metabolic lesion of the brain, even without a history of seizure, and without anticonvulsant medication
7. History of seizures or epilepsy
8. Receiving drugs acting primarily on the central nervous system, which lower the seizure threshold
9. Pregnant females
10. If a woman of childbearing age is unsure of the pregnancy, and does not want to take the pregnancy test
11. Ongoing cord compression or a syrinx in the spinal cord or who suffer from a spinal cord disease such as spinal stenosis, spina bifida, MS, or herniated disk
12. Metal plate in skull
13. Individuals with scalp shrapnel, cochlear implants, or aneurysm clips
14. Individuals taking Bupropion, Dolutegravir, Lacosamide, Trilaciclib, or PR Interval prolonging drugs

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-02-28 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Motor evoked potentials (MEPs) | MEPs measured at baseline, 7 weeks (20 sessions), and 14 weeks (40 sessions) of STDP stimulation and respiratory training for the participants during study procedures.
  Transcranial magnetic stimuli (TMS) will be delivered to the optimal scalp position for activation of the diaphragm muscle. The optimal scalp position will be determined by moving the coil in small steps along the diaphragm representation of the primary motor cortex to find the region where the largest MEP can be evoked with the minimum intensity in the targeted muscles.
Change in Maximum Voluntary Contractions (MVCs) | MVCs measured at baseline, 7 weeks (20 sessions), and 14 weeks (40 sessions) of STDP stimulation and respiratory training for the participants during study procedures.
  Individuals will perform a maximum voluntary contraction (MVC) of diaphragm muscle through surface electrodes secured to the skin over the chest and belly region.

SECONDARY OUTCOMES:
Change in Cervicomedullary electric potentials (CMEPs) | CMEPs measured at baseline, 7 weeks (20 sessions), and 14 weeks (40 sessions) of STDP stimulation and respiratory training for the participants during study procedures.
  Transcranial magnetic stimuli will be delivered to the optimal position of the cervical spine. A small device on the surface of the skin behind the ear will deliver pulses of electricity over the back of the neck.
Change in Pulmonary function tests | Change in pulmonary function tests measured at baseline, 7 weeks (20 sessions), and 14 weeks (40 sessions) of STDP stimulation and respiratory training for the participants during study procedures.
  Spirometry will be tested in upright and supine position to measure negative inspiratory force (NIF), vital capacity (VC), forced vital capacity (FVC), forced expiratory volume in one second (FEV1) and their ration (FEV1/FVC)
Change in the Diaphragm ultrasound imaging | Change in the diaphragm ultrasound imaging measured at baseline, 7 weeks (20 sessions), and 14 weeks (40 sessions) of STDP stimulation and respiratory training for the participants during study procedures.
  Ultrasound imaging will be acquired for optimal visualization of each hemidiaphragm. The diaphragm will be examined during quiet breathing and during maximal inspiration. MVCs measured at baseline, 7 weeks (20 sessions), and 14 weeks (40 sessions) of STDP stimulation and respiratory training for the participants during study procedures.

CONTACTS AND LOCATIONS:
Overall Officials: Monica A Perez, PT, PhD, Principal Investigator — Shirley Ryan AbilityLab
Locations (1):
- Shirley Ryan Ability Lab, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No